CLINICAL TRIAL: NCT00494468
Title: Single Dose Pharmacokinetic and Pharmacodynamic Evaluation of Three Different Zolpidem Doses in Children Ages 2 to 18 Years of Age
Brief Title: Single Dose Pharmacokinetic and Pharmacodynamic Evaluation of Three Different Doses of Zolpidem in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Sanofi-Synthelabo (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPRU-10590
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2007-06-29 (Estimated); Status verified 2005-11

CONDITIONS: Insomnia; Sleep Disorder
Keywords: Insomnia; Sleep Disorder; Sleep Deprivation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Sleep Deprivation | interventions — Zolpidem

INTERVENTIONS:
Drug: Zolpidem

SUMMARY:
This is a multicenter trial to evaluate the single-dose safety, tolerability and pharmacokinetics-pharmacodynamics of Zolpidem in a group of children with sleep disturbances stratified by age and dose.

DETAILED DESCRIPTION:
The consequences of sleep deprivation to the productivity of the individual and society are extensive. (Most clinicians and patients believe that insomnia becomes a clinical problem requiring therapy when excessive daytime sleepiness impairs cognition and mood, interfering with a patient's performance of functions that require alertness. Chronic sleep deprivation often leads to adverse personal, medical and psychiatric complications, underscoring the common request of patients for treatment by their physician.

With an increasing focus on the problem of sleep deprivation in children of all ages, our appreciation of the scope of the problem is expanding. It is estimated that up to 40 % of infants experience difficulty in settling and frequent nighttime wakings with sleep disturbances including bedtime resistance, delayed onset of sleep, and disruptive night wakings occurring in 25 to 50 % of preschoolers. In school-aged children, parents reported an incidence of bedtime resistance in 15 % of their children.

Very limited data exist describing the pharmacokinetics of zolpidem in pediatrics. Colle and colleagues reported the zolpidem clearance to be 3 times greater in children (n=6) compared to young adults (n=104) though Cmax and AUC values were similar despite a higher zolpidem dose (mg/Kg) in the children. Unfortunately these data raise more questions than they answer regarding zolpidem disposition relative to age and highlight the need to comprehensively determine zolpidem disposition characteristics across a broad age range of pediatric subjects.

In summary, although researchers have been hesitant to include children in drug studies, the data indicate that pediatric sleep disturbance have a negative health impact on children and warrant pharmacologic intervention. Studies to identify the appropriate drug and dosage for children of all ages are essential in addressing this health problem that impacts the child and his/her family.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 2 years and 18 years.
2. Written consent must be obtained form the parent/legal guardian for all minors. Written assent must be obtained from all minors > 6 years of age.
3. Female subjects of child-bearing potential must not be pregnant and if females are fertile and sexually active, must have documented a negative urine HCG and assure use of effective contraception acceptable to the investigator (abstinence accepted) during the study period.
4. Subjects must meet the following criteria for a diagnosis of insomnia as determined by the subject's private physician or study investigator and subject's history:

   * the complaint is significant difficulty (defined by frequency, severity, and/or chronicity) initiating or maintaining sleep;. The problem is viewed problematic by the child and/or caregiver;
   * the sleep disturbance causes clinically significant impairment in school performance, behavior, learning, or development for the child as reported by the child and/or caregiver;
   * the sleep disturbance does not occur exclusively in the context of an intrinsic dyssomnia such as narcolepsy, restless legs syndrome, or sleep-related breathing disorders; a circadian rhythm disorder; or a parasomnia;
   * the sleep disturbance is not attributable to either the direct physiologic effect of a drug of abuse or misuse of a prescribed medication.

Exclusion Criteria:

1. Pregnancy and/or breastfeeding;
2. The presence of any untreated (where treatment is available), or unstable, progressive, or evolving clinically significant renal, endocrine, hepatic, respiratory, cardiovascular, neurologic, hematologic, immunologic, cerebrovascular disease or malignancy;
3. Elevations in screening blood tests of renal (SCr) and liver (ALT, AST and/or bilirubin) > 2 times the upper limit of normal for age.
4. Receiving any medications that may modulate Zolpidem metabolism, primarily drugs that will enhance or reduce the activity of CYP450 3A, 2C9, or 2D6 activity. Note: If patient is receiving a medication that might be considered an inducer or an inhibitor, please discuss with the PI prior to excluding them.
5. Receiving any medications with sleep-impairing properties at a dose/dose interval that would be judged by the study investigator as to interfere with the assessment of Zolpidem sleep response.
6. Currently using any systemic contraceptive steroids including: oral contraceptives, transdermal patch, vaginal insert, levonorgestrel implant and medroxyprogesterone acetate contraceptive injection.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63
Dates: Start 2002-10; Study Completion 2004-03

PRIMARY OUTCOMES:
Safety will be assessed by collection of reported adverse events or findings on physical examination or laboratory assessments.
The primary pharmacokinetic outcome measures for this study will include the Zolpidem Cmax, Tmax, t1/2, AUC (zero to 12 hours and zero to infinity).
Polysomnography, including an electroencephalogram, electrooculogram and electromyogram will be performed on two occasions and represents the primary pharmacodynamic outcome assessment for this study.
Measures will include:
Global sleep parameters: time to sleep, total sleep time, duration of sleep period, sleep efficiency, frequency of shifts between sleep stages and number and duration of awakenings
Sleep Latencies; sleep onset latency, Rapid Eye Movement, (REM) latency, slow-wave sleep,(SWS) latency
Sleep Stages (as absolute and relative proportions thereof: sleep stages I, II, III and IV; sleep stage REM; stage awake
Non-Rem/REM Cycle Parameters: duration of the cycles, REM sleep per cycle, SWS sleep per cycle, number of cycles;
Pharmacodynamic outcomes also will be assessed using activity-based monitoring or actigraphy. This technique has demonstrated ability to measure dose-related effects of hypnotics.

SECONDARY OUTCOMES:
Secondary outcome pharmacokinetic outcome measures will include estimation of the apparent Zolpidem Vd/F and CI/F.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L. Blumer, Ph.D., M. D., Principal Investigator — Rainbow Babies and Children's Hospital
Locations (11):
- United States (11):
  - Arkansas Children's Hospital Research Center Inc., Little Rock, Arkansas
  - University of California at San Diego, La Jolla, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Children's Mercy Hospital & Clinics, Kansas City, Missouri
  - Children's Hospital Research Foundation, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Tennessee College of Medicine, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas